The concurrent validity will be analyzed using the Spearman correlation coefficient by correlating the total score of the BESTest with the scores obtained with the Fall Efficiency Scale, the Berg balance scale and the walk and stand test. The same procedure will be carried out for the mini BESTEST. Statistical analysis of the data will be performed using statistical program Statistica.